CLINICAL TRIAL: NCT00538642
Title: Improving Diabetes Risk Factors in Persons With Schizophrenia or Bipolar Disorder by Switching to Ziprasidone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Alexander L. Miller, Principal Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000000010002968; 124932
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
Keywords: schizophrenia; antipsychotics; diabetes; bipolar disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Diabetes Mellitus | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stay on current antipsychotic (No Intervention): Subjects stay on same daily oral antipsychotic treatment as at baseline. Dose adjustments allowable as clinically indicated.
- ziprasidone treatment (Active Comparator): Subjects switch to daily oral ziprasidone from current antipsychotic(s). Dose titrated to clinically effective level.
  Interventions: Drug: ziprasidone

INTERVENTIONS:
Drug: ziprasidone — Patients assigned to ziprasidone arm are cross-titrated from current antipsychotic
  Other Names: Geodon
  Arms: ziprasidone treatment

SUMMARY:
Having a diagnosis of schizophrenia or bipolar disorder and being treated with certain of the newer antipsychotics are risk factors for development of diabetes. Subjects with these risk factors plus obesity and/or family history of diabetes who agree to study participation will undergo an oral glucose tolerance test. If the oral glucose tolerance test demonstrates that the subject is pre-diabetic (elevated glucose levels, but below the diabetic range), he/she will have his/her insulin resistance level measured, prior to random assignment to either stay on current antipsychotic medication or switch to ziprasidone. Insulin resistance will be measured again after four months. The primary hypothesis is that insulin resistance will decrease in those switched to ziprasidone relative to those continuing on their same antipsychotic medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder or bipolar disorder
* BMI>29.9 or family history of diabetes and/or abdominal circumference greater than 88 cm in women or 102 cm in men
* Pre-diabetic oral glucose tolerance test
* Current treatment with olanzapine, risperidone, paliperidone, or quetiapine, or combination of these
* Willing to switch to ziprasidone
* No psychiatric hospitalizations in past three months and judged by treating clinician to be suitable for antipsychotic medication switch
* Able to give informed consent to study

Exclusion Criteria:

* Judged to be currently suicidal, homicidal, or unable to cooperate with treatment
* Unstable serious medical illness
* Current use of drugs that interfere with glucose and fat metabolism (sulfonylureas, metformin, thiazolidinediones). The use of "statins" and fibrates will be allowed ONLY if stable dose for past 3 months.
* Current diagnosis of diabetes
* Fasting blood glucose >125 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-08; Primary Completion 2011-04 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALEXANDER L MILLER, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center At San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Stay on Current Antipsychotic: Subjects stay on same antipsychotic treatment as at baseline.
- Ziprasidone Treatment: Subjects switch to ziprasidone from current antipsychotic(s)
Period: Overall Study
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Started | 10 | 14
Completed | 9 | 9
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment | Total
Number analyzed (Participants) | 10 | 14 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 14 | 24
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.6 (9.05) | 41.43 (8.46) | 40.25 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 14 | 24

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Euglycemic clamp method
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg glucose/kg.min/μIU insulin
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mg glucose/kg.min/μIU insulin | 5.55 (3.51) | 1.88 (1.08)
Statistical Analysis 1: Comparison: Stay on Current Antipsychotic vs Ziprasidone Treatment; Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: Body Mass Index
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
Kg/m2 | 38.4 (10.5) | 39.0 (4.1)

3. Secondary Outcome: Body Mass Index
Time Frame: 4-5 months
Measure: Mean (Standard Deviation); unit: Kg/m2
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
Kg/m2 | 36.0 (6.4) | 38.8 (4.2)

4. Secondary Outcome: Abdominal Circumference
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
cm | 115 (20) | 126 (17)

5. Secondary Outcome: Abdominal Circumference
Time Frame: 4-5 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
cm | 115 (19) | 122 (8)

6. Secondary Outcome: Systolic Blood Pressure
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mm Hg | 118 (15) | 121 (13)

7. Secondary Outcome: Systolic Blood Pressure
Time Frame: 4-5 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mm Hg | 123 (15) | 128 (15)

8. Secondary Outcome: Diastolic Blood Pressure
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mm Hg | 81 (10) | 80 (9)

9. Secondary Outcome: Diastolic Blood Pressure
Time Frame: 4-5 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mm Hg | 82 (9) | 81 (13)

10. Secondary Outcome: Triglycerides
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mg/dL | 183 (166) | 227 (154)

11. Secondary Outcome: Triglycerides
Time Frame: 4-5 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mg/dL | 154 (87) | 252 (179)

12. Secondary Outcome: Cholesterol
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mg/dL | 176 (53) | 176 (36)

13. Secondary Outcome: Cholesterol
Time Frame: 4-5 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mg/dL | 177 (34) | 186 (44)

14. Secondary Outcome: HDL Cholesterol
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mg/dL | 34 (8) | 35 (5)

15. Secondary Outcome: HDL Cholesterol
Time Frame: 4-5 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mg/dL | 40 (9) | 38 (9)

16. Secondary Outcome: LDL Cholesterol
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mg/dL | 108 (43) | 106 (35)

17. Secondary Outcome: LDL Cholesterol
Time Frame: 4-5 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mg/dL | 106 (29) | 109 (35)

18. Primary Outcome: Insulin Sensitivity
Description: Euglycemic clamp method
Time Frame: 4-5 months
Measure: Mean (Standard Deviation); unit: mg glucose/kg.min/μIU insulin
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Number analyzed (Participants) | 9 | 9
mg glucose/kg.min/μIU insulin | 6.01 (3.93) | 2.07 (1.15)

ADVERSE EVENTS:
Arm/Group | Stay on Current Antipsychotic | Ziprasidone Treatment
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/14
Other Adverse Events (participants affected / at risk) | 0/10 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less